CLINICAL TRIAL: NCT00547352
Title: Switching From Sildenafil Citrate to Tadalafil in Treatment of Erectile Dysfunction: Assessment of Treatment Preference
Brief Title: Study to Determine a Preference Between Sildenafil or Tadalafil Treatment for Problems Getting an Erection
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: ICOS Corporation (Industry)
Model: Crossover | Masking: None
Other Study IDs: 9152; H6D-KL-S002
Record Dates: First submitted 2007-10-18; First posted 2007-10-22 (Estimated); Last update posted 2007-10-22 (Estimated); Status verified 2007-10

CONDITIONS: Impotence
MeSH Terms: conditions — Erectile Dysfunction | interventions — Tadalafil; Sildenafil Citrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): sildenafil treatment for at least 10 weeks prior to a 1 week wash out
  Interventions: Drug: sildenafil
- 2 (Active Comparator): Tadalafil treatment for 8 weeks following the 1 week washout period.
  Interventions: Drug: tadalafil

INTERVENTIONS:
Drug: tadalafil — 20 mg tadalafil tablets taken by mouth, as needed, no more than once a day for 8 weeks.
  Other Names: LY450190; Cialis; IC351
  Arms: 2
Drug: sildenafil — Current users of sildenafil citrate for a minimum of 6 weeks prior to visit 1 will continue with an individual dosage to be taken no more than once a day for an additional 4 weeks.
  Arms: 1

SUMMARY:
To determine if men with problems getting and keeping an erection prefer treatment with tadalafil or sildenafil.

ELIGIBILITY:
Inclusion Criteria:

* History of erection problems
* Anticipate a monogamous female sexual relationship
* Abstain from other erection treatments throughout the study
* Currently use sildenafil

Exclusion Criteria:

* Other primary sexual disorders
* History of radical prostatectomy or other pelvic surgery that affected being able to have an erection
* History of penile implant or clinically significant penile deformity.
* Nitrate use
* Certain heart problems

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2004-06; Study Completion 2005-06 (Actual)

PRIMARY OUTCOMES:
Patient choice of drug at visit 5 | 14-15 weeks

SECONDARY OUTCOMES:
PAIRS self-administered scale scores | 14-15 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon- Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Seoul, South Korea

REFERENCES:
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com